CLINICAL TRIAL: NCT00112073
Title: A Phase IIA, Multicenter, Randomized, Double-Blind, Placebo-Controlled, Multiple Ascending Dose, Safety, Tolerability, Pharmacokinetic, Pharmacodynamic, and Immunogenicity Trial of AAB-001 in Patients With Mild to Moderate AD
Brief Title: AAB-001 in Patients With Mild to Moderate Alzheimer's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: JANSSEN Alzheimer Immunotherapy Research & Development, LLC (Industry)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AAB-001-201
Record Dates: First submitted 2005-05-27; First posted 2005-05-30 (Estimated); Last update posted 2012-03-14 (Estimated); Status verified 2012-03

CONDITIONS: Alzheimer's Disease
Keywords: Alzheimer's disease; immunotherapy; beta amyloid
MeSH Terms: conditions — Alzheimer Disease; Plaque, Amyloid | interventions — bapineuzumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (8):
- 0.15 mg/kg active bapineuzumab (Experimental)
  Interventions: Drug: bapineuzumab
- 0.15 mg/kg placebo (Placebo Comparator)
  Interventions: Other: placebo
- 0.5 mg/kg active bapineuzumab (Experimental)
  Interventions: Drug: bapineuzumab
- 0.5 mg/kg placebo (Placebo Comparator)
  Interventions: Other: placebo
- 1.0 mg/kg active bapineuzumab (Experimental)
  Interventions: Drug: bapineuzumab
- 1.0 mg/kg placebo (Placebo Comparator)
  Interventions: Other: placebo
- 2.0 mg/kg active bapineuzumab (Experimental)
  Interventions: Drug: bapineuzumab
- 2.0 mg/kg placebo (Placebo Comparator)
  Interventions: Other: placebo

INTERVENTIONS:
Drug: bapineuzumab — IV, Q13w
  Other Names: AAB-001
  Arms: 0.15 mg/kg active bapineuzumab; 0.5 mg/kg active bapineuzumab; 1.0 mg/kg active bapineuzumab; 2.0 mg/kg active bapineuzumab
Other: placebo — IV Q13w
  Arms: 0.15 mg/kg placebo; 0.5 mg/kg placebo; 1.0 mg/kg placebo; 2.0 mg/kg placebo

SUMMARY:
The purpose of this study is to assess the safety and tolerability of multiple doses of AAB-001 passive immunization in patients with mild to moderate Alzheimer's disease (AD).

DETAILED DESCRIPTION:
The humanized monoclonal antibody, AAB-001, which binds to and clears beta amyloid peptide, is designed to provide antibodies to beta amyloid directly to the patient, rather than requiring the patient to mount his/her own individual response. It is believed that this approach may eliminate the need for the patient to mount an immune response to beta amyloid. Animal studies have shown that this approach is equally effective in clearing beta amyloid from the brain as traditional active immunization methods.

This is a multicenter, double-blind, placebo controlled, randomized, outpatient, multiple ascending dose study in male and female patients aged 50 to 85 years with mild to moderate AD. Approximately 30 study sites will be involved. Patients will be randomized to receive either AAB-001 or placebo. Each patient's participation will last approximately 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of probable AD
* Age from 50 to 85 years
* Rosen Modified Hachinski Ischemic score less than or equal to 4
* Magnetic resonance imaging (MRI) scan consistent with the diagnosis of AD
* Fluency in English
* Stable doses of medications

Exclusion Criteria:

* Significant neurological disease other than AD
* Major psychiatric disorder
* Significant systemic illness
* History of stroke or seizure
* Weight greater than 120 kg (264 lbs.)
* History of autoimmune disease
* Smoking more than 20 cigarettes per day
* Anticonvulsants, anti-Parkinson's, anticoagulant, or narcotic medications
* Prior treatment with experimental immunotherapeutics or vaccines for AD
* Presence of pacemakers or foreign metal objects in the eyes, skin, or body

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 234 (Actual)
Dates: Start 2005-04; Primary Completion 2008-11 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
safety assessments | 18 months

SECONDARY OUTCOMES:
blood levels of administered study drug | 18 months
cognitive and functional assessments | 18 months

CONTACTS AND LOCATIONS:
Locations (26):
- United States (26):
  - Cleo Roberts Center for Clinical Research / Sun Health Research Institute, Sun City, Arizona
  - UC Irvine, Irvine, California
  - Pharmacology Research Institute, Los Alamitos, California
  - Pharmacology Research Institute, Northridge, California
  - UCSD Shiley-Marcos Alzheimer's Disease Research Center, San Diego, California
  - Memory & Aging Center, UCSF, San Francisco, California
  - Yale University School of Medicine, New Haven, Connecticut
  - Georgetown University Medical Center, Washington D.C., District of Columbia
  - Brain Matters Research, Inc., Delray Beach, Florida
  - Mayo Clinic - Department of Neurology, Jacksonville, Florida
  - Rush Presbyterian St. Luke's Medical Center, Chicago, Illinois
  - Department of Neurology - Indiana University Medical Center, Indianapolis, Indiana
  - Behavioral Neurology, Boston, Massachusetts
  - University of Michigan Health System, Department of Neurology, Ann Arbor, Michigan
  - Mayo Clinic Department of Neurology - Alzheimer's Disease Research Center, Rochester, Minnesota
  - The Memory Enhancement Center, Long Branch, New Jersey
  - Sergievsky Center, Columbia University, New York, New York
  - University of Rochester / Monroe Community Hospital, Rochester, New York
  - Department of Psychiatry and Behavioral Sciences, Durham, North Carolina
  - Oregon Health and Science University, Portland, Oregon
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Memory and Aging Program, Butler Hospital, Providence, Rhode Island
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Baylor College of Medicine, Houston, Texas
  - Clinical Neuroscience Research Associates, Inc., Bennington, Vermont
  - University of Washington, Seattle, Washington

REFERENCES:
- [Derived] Arrighi HM, Barakos J, Barkhof F, Tampieri D, Jack C Jr, Melancon D, Morris K, Ketter N, Liu E, Brashear HR. Amyloid-related imaging abnormalities-haemosiderin (ARIA-H) in patients with Alzheimer's disease treated with bapineuzumab: a historical, prospective secondary analysis. J Neurol Neurosurg Psychiatry. 2016 Jan;87(1):106-12. doi: 10.1136/jnnp-2014-309493. Epub 2015 Feb 10. PMID 25669746
- [Derived] Blennow K, Zetterberg H, Rinne JO, Salloway S, Wei J, Black R, Grundman M, Liu E; AAB-001 201/202 Investigators. Effect of immunotherapy with bapineuzumab on cerebrospinal fluid biomarker levels in patients with mild to moderate Alzheimer disease. Arch Neurol. 2012 Aug;69(8):1002-10. doi: 10.1001/archneurol.2012.90. PMID 22473769